CLINICAL TRIAL: NCT03083977
Title: Examining the Effects of Processed Music on Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pandemic related difficulties for recruitment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephen Porges, Distinguished University Scientist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1702490842
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): This group will listen to 1 hour of processed music (Safe and Sound Protocol) for 5 days
  Interventions: Other: Safe and Sound Protocol

INTERVENTIONS:
Other: Safe and Sound Protocol — The intervention features music processed based on the resonating frequencies of the middle ear

SUMMARY:
Chronic pain is a common ailment in aging populations and often co-occurs with altered regulation of the autonomic nervous system. Nociceptive pathways (i.e., those that transmit pain signals) are integrated with autonomic circuits throughout the body and therapies that are successful in reducing pain concurrently alter autonomic functions, even when they are not directly designed to do so. It is possible that interventions that target the autonomic circuits that regulate pain responses may help reduce pain in chronic pain sufferers. The proposed study will examine whether an intervention that targets the autonomic nervous system via filtered music can reduce pain, a hypothesis derived from the Polyvagal Theory.

The Polyvagal Theory describes how function and structure of the vertebrate autonomic nervous system changed during evolution. The theory is named for the vagus, a major cranial nerve that regulates bodily state. An evolutionary "old" branch of this nerve innervates structures below the diaphragm and its dysfunction is linked to lower body organ and tissue pain. Regulation of the vagus nerve is linked with specific auditory cues based on our evolutionary heritage and the physics of the middle ear. This study is designed to test whether processed music designed to stimulate vagal function can decrease chronic pain. The Listening Project Protocol, the processed music used in this intervention, has previously been shown to effectively stimulate the function of the vagus nerve (see stimulus description below).

Specific Aims:

Aim I: To examine whether The Listening Project Protocol, a non-invasive audio intervention, can be effective for reducing chronic pain in a sample of older adults.

Hypothesis: Five 1-hour sessions of the Listening Project Protocol will reduce pain

Aim II: To examine whether increased regulation via the autonomic nervous system accounts for the decrease in pain if the intervention is successful.

Hypothesis: Pain reduction will coincide with improved autonomic function by the myelinated vagus nerve (measured by respiratory sinus arrhythmia, see below) as well as decrease in the reactivity of autonomic functions in everyday experiences (measured by the Body Perception Questionnaire, see below)

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-report as suffering from chronic pain

Exclusion Criteria:

* Individuals who do not read or speak proficient English
* Individuals with substantial, uncorrected hearing loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change over 1 week
  Change in intensity of pain from pre-assessment to post-assessment, measured by the Brief Pain Inventory Short Form
Pain experience | Change over 1 week
  Change in experience of pain from pre-assessment to post-assessment, measured by the McGill Pain Questionnaire Short Form

SECONDARY OUTCOMES:
Autonomic Function | Change over 1 week
  Amplitude of respiratory sinus arrhythmia (RSA), a measure of myelinated vagal effects on the heart
Body perception | Change over 1 week
  Autonomically-mediated body perception, measured by the Body Perception Questionnaire Short Form

OTHER OUTCOMES:
Auditory processing | Change over 1 week
  Auditory speech processing measured by ability to extract speech from background noise and understand speech with frequencies removed; measured by the SCAN Test for Auditory Processing Disorders (Keith, 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Porges, PhD, Principal Investigator — Indiana University; Peter Miksza, PhD, Study Chair — Indiana University; Hannah Fidler, Study Chair — Indiana University; Jacek Kolacz, PhD, Study Chair — Indiana University
Locations (1):
- Meadowood Retirement Community, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No